CLINICAL TRIAL: NCT06562647
Title: An Exploratory Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics, and Initial Efficacy of SY001 Injection Targets Mesothelin in a Single-arm, Dose-increasing Setting in Subjects With Advanced Solid Tumors
Brief Title: SY001 Targets Mesothelin in a Single-arm, Dose-increasing Setting in Subjects With Advanced Solid Tumors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cell Origin Biotech (Hangzhou) Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Xudong Wang, manager, Cell Origin Biotech (Hangzhou) Co., Ltd.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2303
Record Dates: First submitted 2024-08-15; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Treatment Related Cancer; Ovarian Cancer
MeSH Terms: conditions — Neoplasms, Second Primary; Ovarian Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SY001 Targets Mesothelin positive solid tumors in a Dose-increasing Setting (Experimental): Patients with mesothelin-positive ovarian cancer were treated with an SY001 injection in combination with an anti-PD-1 antibody. Patient 001 received 1109 SY001 CAR-pMACs via intravenous injection. Following a two-month period in which the treatment's safety was confirmed, this patient underwent another two does of 1109 SY001 cells on both day 1 and day 3. Prior to the CAR-pMACs infusion on day 1, a PD1 antibody Tislelizumab Injection was administered. In the case of the patient 002, SY001 treatment was delivered intravenously on three occasions: day 1, day 3, and day 5. The same as the first patient's protocol, Tislelizumab was given prior to the CAR-pMACs on day 1.
  Interventions: Drug: SY001

INTERVENTIONS:
Drug: SY001 — PBMC-derived anti-mesothelin Cheimeric Antigen Receptor macrophages
  Other Names: CAR-pMAC

SUMMARY:
Single-arm, dose-increasing setting study of CAR macrophages in Mesothelin overexpressing solid tumors.

DETAILED DESCRIPTION:
This study was a single-arm, single-center, dose-increasing design, using the "3+3" approach for dose escalation, to evaluate the safety, tolerability and initial effectiveness of SY001, and to evaluate the pharmacokinetic characteristics, cytokines and the correlation between the efficacy of SY001.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pathologically diagnosed advanced ovarian cancer/pancreatic cancer who have failed at least 1 prior lines treatment, and tumor tissue samples were positive for mesothlin IHC staining;
2. According to the RECIST 1.1, there is measurable tumor lesions (non-lymph node lesion 10mm in length or lymph node lesion 15mm in diameter measured by CT or MRI, with scan layer thickness 5mm);
3. Eastern Cooperative Oncology Group (ECOG) score of 2 and satisfactory major organ functions;
4. Estimated life expectancy >3 months;
5. Female patients of childbearing age must undergo a serum pregnancy test at screening and prior to pretreatment and the results must be negative, and are willing to use a very effective and reliable method of contraception within 1 year after the last study treatment.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Any uncontrollable active infection, including but not limited to active tuberculosis, HBV infection;
3. Patients who have a history of other mesothelin-targeting therapy;
4. Patients who have a history of autoimmune disease;
5. The investigator assessed that the patient was unable or unwilling to comply with the requirements of the study protocol.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Identification of Maximum Tolerated Dose (MTD) | up to 28 days after SY001 infusion.
  MTD will be determined based on DLTs observed during the first 28 days of study treatment.

SECONDARY OUTCOMES:
Objective response rate (ORR) | 3 months
  Treatment response was assessed according to the criteria of RECIST 1.1, with PET-CT scans being the primary method used to evaluate tumor progression.
Time to Peak (Tmax) | 1 month
  Changes in the CAR gene copy number after infusion of SY001; time to peak (Tmax) from 0 to 1 month.
Area Under the Plasma Concentration Versus Time Curve (AUC) | 1 month
  Changes in the CAR gene copy number after infusion of SY001, area under the concentration-time curve (AUC) from 0 to 1 month
Maximum Plasma Concentration of cytokines (Cmax) | 1 month
  Changes in cytokines in peripheral blood after infusion of SY001.

CONTACTS AND LOCATIONS:
Locations (1):
- Linyi Cancer Hospital, Linyi, China